CLINICAL TRIAL: NCT05294471
Title: Fully Automated High-Throughput Quantitative MRI of the Liver
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-1615; 2021-1615 (Other: UW Madison); A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); 4/29/2025 (Other: UW Madison); 1R01EB031886-01A1 (NIH)
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Iron Overload; Liver Fat
MeSH Terms: conditions — Iron Overload; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Healthy participants: 70 healthy participants will be recruited, across substudies 1, 2, 4, and 5
  Interventions: Device: Non-contrast MRI with novel MRI software
- Participants with known or suspected iron overload: 30 Participants with known or suspected iron overload will be recruited, to substudy 3
  Interventions: Device: Non-contrast MRI with novel MRI software
- Participants with elevated levels of liver fat: 30 participants with elevated levels of liver fat will be recruited, to substudy 3
  Interventions: Device: Non-contrast MRI with novel MRI software
- Participants referred for clinical abdominal MRI: 60 participants referred for clinical abdominal MRI will be recruited, to substudy 6
  Interventions: Device: Non-contrast MRI with novel MRI software

INTERVENTIONS:
Device: Non-contrast MRI with novel MRI software — The investigational software being used in automatic prescription of the imaging is an application of an AI algorithm. This software prescribes where the MRI system will take images by finding the liver within a set of localizer scans. The software gives coordinates to the scanner.

SUMMARY:
The purpose of this research is to see if a new automated magnetic resonance imaging (MRI) method will be able to improve the images taken of the liver. Participants will have either known or suspected liver disease, known or suspected iron overload syndrome, or be a healthy adult. Participants will be in the research study for one day.

DETAILED DESCRIPTION:
The overall purpose of this work is to develop, implement and test a "single-button push", integrated combination of innovative MRI solutions to enable low-cost quantitative evaluation of chronic liver disease in less than 5 minutes of true MRI suite time. The aim is to design a reliable, low variability, fully automated, highly efficient MRI exam.

The primary objective is to demonstrate a free-breathing 2D CSE-MRI method that is robust to motion and free of bias when compared to the reference 3D CSE-MRI method.

Secondary objectives include optimization of the methods in healthy volunteers, and technical success and throughput of the single-button push exam:

1. Repeatability: we will calculate the squared difference between each pair of repeated proton density fat fraction (PDFF) / R2* measurements, and will model this value including the acquisition/reconstruction method as a covariate using Generalized Estimating Equations (GEE)
2. Reproducibility of the proposed method between 1.5T and 3T using the reproducibility coefficient and interclass correlation coefficient (ICC)
3. Technical success of the single-push button exam (completion of exam, acceptable automated prescription as determined through radiologist evaluation, image quality, and automated analysis accuracy compared to manual analysis)
4. Mean and standard deviation of total two-door suite time for the single-push button exam

Specific Aims:

Aim 1: Develop and optimize motion-insensitive, high-SNR (signal-to-noise ratio), free-breathing "error-proof" CSE-MRI for accurate and precise measurement of PDFF and R2* as biomarkers of liver fat and iron.

Aim 2: Confirm the accuracy (ie: bias) and precision (ie: repeatability, and reproducibility across field strength) of the proposed CSE-MRI method in patients with liver steatosis and in patients with liver iron overload.

Aim 3: Implement and validate an integrated single-button push, fully automated CSE-MRI protocol in < 5 minutes of MR room time, using i) Artificial intelligence (AI)-based automated image prescription, ii) an innovative MRI "Smart Suite" design, and iii) automated quantitative image analysis and reporting.

To accomplish these aims, participants will be recruited for 6 substudies:

1. Substudy 1: Optimization of free breathing 2D CSE method in healthy volunteers
2. Substudy 2: Validation of free breathing 2D CSE method in healthy volunteers
3. Substudy 3: Validation in patients with known or suspected iron overload or fatty liver
4. Substudy 4: Evaluation of auto-prescription in healthy volunteers
5. Substudy 5: Round-robin evaluation of single-push button exam in healthy volunteers
6. Substudy 6: Throughput evaluation in patients scheduled for clinical abdominal MRI

For substudies 1, 2, and 4 participants will be asked to complete one research visit lasting approximately 1.5 hours. Participants will be scanned at a single field strength for up to 1 hour. To assess test-retest repeatability, subjects may be asked to sit up on the MRI scanner bed, or step off then back on to the scanner.

In substudy 3, participants will be asked to complete one research visit lasting approximately 1.5 hours. Participants will be scanned on a 1.5T system for up to 1 hour. In order to demonstrate the reproducibility across field strength of CSE MRI to measure liver iron and fat, 10 participants with liver fat and 10 participants with liver iron will be scanned a second time on the same day at 3T. For these 20 participants, total scan time be less than 2 hours and the study visit will last approximately 3 hours.

In substudy 5, the study visit will last approximately 3.5 hours. Participants will participate in groups of 10. After consenting, MRI screening, and anthropometric measurements, participants will form a queue and be scanned consecutively. After scanning, each participant will rejoin the end of the queue. Each participant will be scanned 3 times. Each individual scanning "session" will last approximately 5 minutes, and each participants total scan time will be less than 20 minutes.

Each participant in substudy 5 will be equipped with a Smart Suite RFID (radio frequency identification) or Bluetooth bracelet system to track MRI suite time for each participant and scan. The bracelets are also used in clinical imaging visits to track patient workflow. The bracelet will be used to track when participants enter and leave the MRI suite. The relative timings from baseline will be recorded automatically, entered into the study RedCap and linked with other study data via the participant's Study ID.

For substudy 6, prior to their clinical exam, participants will be scanned with the single-button push protocol. The research scan time will be less than 10 minutes and the total research visit will last approximately 20 minutes. Each participant in this substudy will also be equipped with a Smart Suite RFID or Bluetooth bracelet system to track MRI suite time for each participant and scan, as described for substudy 5.

ELIGIBILITY:
Eligibility Criteria for Substudies 1, 2, 4, 5

Inclusion Criteria:

* Age 18 years or older

Exclusion Criteria:

* Patients with contraindication to MRI (e.g. pacemaker, contraindicated metallic implants, claustrophobia, etc)
* Pregnant or trying to become pregnant (as determined by self-report during MRI safety screening)

Eligibility Criteria for Substudy 3

Inclusion Criteria:

* Age 7 years or older
* One of:

  * Known or suspected liver iron overload
  * Known or suspected elevated liver fat

Exclusion Criteria:

* Patients with contraindication to MRI (e.g. pacemaker, contraindicated metallic implants, claustrophobia, etc)
* Sedation required for MRI
* Pregnant or trying to become pregnant (as determined by self-report during MRI safety screening)

Eligibility Criteria for Substudy 6

Inclusion Criteria:

* Age 7 years or older
* Scheduled for a clinical abdominal MRI exam

Exclusion Criteria:

* Patients with contraindication to MRI (e.g. pacemaker, contraindicated metallic implants, claustrophobia, etc)
* Sedation required for MRI
* Pregnant or trying to become pregnant (as determined by self-report during MRI safety screening)

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers will be recruited from the "MRI Volunteer Database", and/or UW - Madison employees.
  Participants with liver fat or liver iron will be recruited from relevant UW Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Confirm the accuracy (ie: bias) of the proposed CSE-MRI method in patients with liver steatosis and in patients with liver iron overload | 1 day (1 study visit, up to 3.5 hours)
  For each liver segment, and for whole-liver PDFF and R2* measurements, we will determine bias of CSE 2D using CSE 3D BH as the reference from Bland-Altman analysis.
  The range of R2* values leading to reliable measurements of PDFF and R2* will be determined using a two-segment piecewise linear model with the change point estimated from the data.

SECONDARY OUTCOMES:
Image quality of free breathing 2D chemical shift encoded (CSE) method | 1 day (1 study visit, up to 3.5 hours)
  Image quality for each acquisition will be evaluated by 3 radiologists, using a Likert scale between 0 (worst/non-diagnostic) and 3 (best) for criteria including: motion artifacts, spatial resolution, SNR (signal- to-noise ratio), and overall image quality.
Measure the repeatability of the proposed CSE-MRI method in patients with liver steatosis and in patients with liver iron overload | 1 day (1 study visit, up to 3.5 hours)
  To compare repeatability for various acquisition/reconstruction methods, we will calculate the squared difference between each pair of repeated PDFF / R2* measurements, and will model this value including the acquisition/reconstruction method as a covariate using Generalized Estimating Equations (GEE), with subject as a random factor to account for within-subject correlation. This analysis will be performed for all liver segments and whole-liver measurements. Further, the repeatability coefficient will also be assessed separately for each method. Bland-Altman plots will also be used to visualize the repeatability profile over the PDFF / R2* range. The automated vs manual PDFF / R2* measurements will be evaluated for each acquisition.
Confirm the reproducibility of the proposed CSE-MRI method across field strengths | 1 day (1 study visit, up to 3.5 hours)
  The reproducibility of the proposed method between 1.5T and 3T will be evaluated in two ways. First, at each field strength, PDFF and R2* will each be compared between FB FAM CSE and BH CSE 3D (as the reference), using Bland Altman analysis to assess the bias. Second, PDFF will be compared between 1.5T and 3T using Bland Altman analysis for each method, based on the expected field strength independence of PDFF. R2* will also be compared between 1.5T and 3T for each method, after converting to liver iron concentration (LIC, mg/g) using the 1.5T and 3T calibrations determined by our group, to compensate for the effect of field strength on R2*. In all comparisons, the reproducibility coefficient, and interclass correlation coefficient (ICC) with 95% confidence intervals will be calculated to quantify the degree of reproducibility.
Technical success rate of the integrated single-button push, fully automated CSE-MRI protocol in < 5 minutes of MR room time | 1 day (1 study visit, up to 3.5 hours)
  The technical success rate of the integrated single-button push, fully automated CSE-MRI exam will be determined through completion rate of the exam in less than 5 minutes, radiologist evaluation of image quality using a Likert scale, and accuracy of the automated analysis compared to manual evaluation.
Mean and standard deviation of total two-door suite time for the single-push button exam | 1 day (1 study visit, up to 3.5 hours)
  Throughput of the single-button push exam will be quantified by: throughput (subjects/hour), suite time per subject (mean, standard deviation, median, and quartiles) and suite time components (eg: room turnaround time, prescan/scan time for each series).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reeder, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes